CLINICAL TRIAL: NCT06170320
Title: STREngthening Epidemiological Surveillance in Benin and Burkina Faso for an Effective Response to COVID-19
Brief Title: STREngthening COronavirus Disease 2019 (COVID-19) Surveillance in Africa
Acronym: STREESCO
Status: Completed | Type: Observational
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Institut de Recherche Clinique du Bénin (Unknown); Barcelona Institute for Global Health (Other); Ministère de la Santé - Bénin (Unknown); Ministère de la Santé et de Hygiène Publique - Burkina Faso (Unknown)
Responsible Party: Sponsor
Other Study IDs: RIA2020EF-2923
Record Dates: First submitted 2023-12-12; First posted 2023-12-14 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: COVID-19; SARS CoV 2 Infection; COVID-19 Pandemic
Keywords: COVID-19; Epidemiological surveillance; Benin; strategic sites; dynamics
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this observational study was to develop, with the intended users, an epidemic surveillance and response system that will be effective, sensitive, coordinated and appropriate.

The STREESCO project aims to

* Implement active epidemiological surveillance of suspected cases in Benin at strategic sites in accordance with the World Health Organization (WHO) protocol, in support of the national strategy for responding to the CoVID-19 virus.
* To strengthen this national strategy by developing a clinico-epidemiological surveillance system in remote areas of Benin (health centre approach) and Burkina Faso (population survey approach).
* To gain a better understanding of the dynamics of the epidemic and its parameters in Africa thanks to a modern biostatistical and geo-epidemiological analysis of the data collected as part of this project.

DETAILED DESCRIPTION:
Within the framework of the health systems set up by the Benin health authorities, the project aims to develop, with the intended users, an epidemic surveillance and response system that will be effective, sensitive, coordinated and adapted to a context where resources are limited. Following the start of data collection on 01 March 2021, new reforms to the response strategy against CoVID-19 in Benin have led the investigators to opt for a new strategy in order to meet the objectives of the study. The epidemiological surveillance system will be adapted to the reforms, and data collected and processed prospectively on the dynamics of the epidemic will be collected in CoVID-19 screening centres and in public and private health centres. This is the scientific data needed to issue an early warning signal and enable the healthcare system to respond appropriately. The information system will be based on (i) epidemiological surveys in the field, (ii) virological, serological and antigenic tests, (iii) indicators that will enable action to be monitored, adaptation to the epidemic to be assessed and the response capacity of health structures to be controlled. Analysis (biostatistics, geo-epidemiology) of the data collected will provide useful knowledge for a better understanding of the dynamics of the epidemic. Finally, the project will encourage collaboration between African and European researchers and strengthen the capacity of African institutions to set up an epidemic surveillance system.

ELIGIBILITY:
Inclusion Criteria:

* All volunteering for COVID-19 screening in health units dedicated to COVID-19 activities.
* Having benefited from a COVID-19 test.
* Give free and informed consent to participate in the study.

Exclusion Criteria:

* Subjects who did not give free and informed consent to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This surveillance was carried out in 03 strategic sites: in Cotonou, the economic capital, in Allada, a town on the border of the cordon sanitaire set up in March 2020, and in Natitingou, a town in northern Benin outside the cordon sanitaire. It was based in the health units involved in the response to COVID-19 at the 03 strategic sites. Initially, we included volunteers for COVID-19 screening, contact cases of positive subjects, and health workers present in the centres. Secondly, The study population consisted of pregnant women in the third trimester (≥ 28 weeks) of pregnancy seen for antenatal care (ANC) in the study maternity units of the 03 strategic sites were surveyed in order to describe their serological status with respect to SARS-CoV-2 infection.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects infected with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) by strategic sites (suspected cases, contact cases) | 9 months
  Total number of subjects with a positive COVID-19 test divided by the total number of volunteers tested in the study.
Average number of contact cases per person infected with SARS-CoV-2 across all the study sites was as follows | 9 months
  Identify the number of contact cases per subject testing positive for SARS-CoV-2 infection at each of the strategic sites.
Factors associated with SARS-CoV-2 infection in volunteers screened at 03 strategic sites | 9 months
  Multivariate logistic regression model on sociodemographic, anthropometric, clinical and environmental characteristics of volunteer subjects screened for SARS-CoV-2 infection
Clusters of cases in the area of each strategic site (radius, period, relative risk) | 9 months
  Analysis of the spatial distribution of positive cases of SARS-CoV-2 infection on each of the strategic sites
Intra-district incidence rate on the 03 strategic sites | 9 months
  Number of positive cases for SARS-CoV-2 infection divided by the total number of the population multiplied by 1000.
Environmental factors associated with incidence rates and hotspots | 9 months
  Binomial mixed generalized additive model (GAMM)
Basic reproduction number for each strategic site and overall | 9 months
  Bayesian approach to quantify transmissibility over time during the epidemic at each site and overall.
Proportion of health workers infected with SARS-CoV-2 by strategic sites | 9 months
  Total number of health workers with a positive COVID-19 test divided by the total number of health workers tested in the study.
Factors associated with SARS-CoV-2 infection in health workers at 03 strategic sites | 9 months
  Multivariate logistic regression model on sociodemographic, anthropometric, clinical and environmental characteristics, prevention and control measures among health workers for SARS-CoV-2 infection.
Seroprevalence of SARS-CoV-2 infection among pregnant women in the 3rd trimester in maternity wards of strategic study sites | 3 months
  Number of pregnant women with a positive Rapid Diagnostic Test (RDT) divided by the total number of pregnant women tested during the study.
Factors associated with SARS-CoV-2 sero-infection in pregnant women in the 3rd trimester at 03 strategic sites | 3 months
  Multivariate logistic regression model on sociodemographic, anthropometric, clinical, linked to the course of pregnancy and vaccination status characteristics in pregnant women in the 3rd trimester at 03 strategic sites

CONTACTS AND LOCATIONS:
Overall Officials: Achille MASSOUGBODJI, Principal Investigator — Institut de Recherche Clinique du Bénin; Gilles COTTRELL, Study Director — Institut de Recherche pour le Développement - France; Raquel GONZALEZ, Study Director — Fundación Privada Instituto de Salud Global Barcelona; Anges YADOULETON, Study Chair — Ministère de la Santé - Bénin; Boukary OUEDRAOGO, Study Chair — Ministère de la Santé - Burkina Faso
Locations (1):
- Institut de Recherche Clinique du Bénin, Abomey-Calavi, Atlantique Department, Benin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atchade A, Yadouleton A, Fiogbe M, Abdoulaye Alfa D, Yovo E, Le Hesran JY, Hounsa S, Bationo C, Figueroa-Romero A, Gaudart J, Gonzalez R, Bonnet E, Massougbodji A, Cottrell G. Determinants of SARS-CoV-2 infection across three sentinels sites in Benin during 2021: A multicentric surveillance study. PLOS Glob Public Health. 2025 Feb 13;5(2):e0004227. doi: 10.1371/journal.pgph.0004227. eCollection 2025. PMID 39946403
- [Derived] Figueroa-Romero A, Atchade A, Yadouleton A, Fiogbe M, Bonnet E, Yovo E, Accrombessi M, Hounsa S, Paper T, Dupont R, Gaudart J, Le Hesran JY, Massougbodji A, Cottrell G, Gonzalez R. SARS-CoV-2 seroprevalence among Beninese pregnant women in the third year of the pandemic. BMC Public Health. 2024 Jul 2;24(1):1762. doi: 10.1186/s12889-024-19087-4. PMID 38956517